CLINICAL TRIAL: NCT00451217
Title: A Multi -Center Randomized Parallel Group Comparative Active Controlled Safety Assessor Blinded Phase 3a Pivotal Trial in Adult Subjects Comparing Org 25969 With Neostigmine as Reversal Agents of a Neuromuscular Block Induced by Rocuronium or Vecuronium at Reappearance of T2
Brief Title: Comparison of Sugammadex (Org 25969) With Neostigmine as Reversal Agents for Rocuronium or Vecuronium at Reappearance of T2 (P05960)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P05960; 19.4.301 (Other: Organon Protocol Number); MK-8616-033 (Other: Merck Protocol Number)
Record Dates: First submitted 2007-03-22; First posted 2007-03-23 (Estimated); Results first posted 2019-02-18 (Actual); Last update posted 2019-03-04 (Actual); Status verified 2019-02

CONDITIONS: Anesthesia, General
MeSH Terms: interventions — Sugammadex; Neostigmine; Glycopyrrolate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Rocuronium + Sugammadex (Experimental): After the last dose of rocuronium, at reappearance of T2, a dose of 2.0 mg/kg sugammadex was administered
  Interventions: Drug: Sugammadex
- Rocuronium + Neostigmine (Active Comparator): After the last dose of rocuronium, at reappearance of T2, a dose of 50 ug/kg neostigmine was administered
  Interventions: Drug: Neostigmine
- Vecuronium + Sugammadex (Experimental): After the last dose of vecuronium, at reappearance of T2, a dose of 2.0 mg/kg sugammadex was administered
  Interventions: Drug: Sugammadex
- Vecuronium + Neostigmine (Active Comparator): After the last dose of vecuronium, at reappearance of T2, a dose of 50 ug/kg neostigmine was administered
  Interventions: Drug: Neostigmine

INTERVENTIONS:
Drug: Sugammadex — After the last dose of rocuronium or vecuronium, at reappearance of T2, a dose of 2.0 mg/kg sugammadex was to be administered
  Other Names: Org 25969
  Arms: Rocuronium + Sugammadex; Vecuronium + Sugammadex
Drug: Neostigmine — After the last dose of rocuronium or vecuronium, at reappearance of T2, a dose of 50 ug/kg neostigmine was to be administered
  Other Names: premix neostigmine/glycopyrrolate
  Arms: Rocuronium + Neostigmine; Vecuronium + Neostigmine

SUMMARY:
The purpose of this study was to demonstrate in adult participants faster recovery from a neuromuscular block induced by either rocuronium or vecuronium after reversal at reappearance of T2 (the amplitude of the first response of second twitch to train of four (TOF) stimulation, expressed as percentage of control first twitch, T1) by 2.0 mg/kg sugammadex (Org 25969) compared to 50 ug/kg neostigmine.

ELIGIBILITY:
Inclusion Criteria:

* Is of American Society of Anesthesiologists (ASA) 1 - 4;
* Is above or equal to the age of 18;
* Scheduled for surgical procedures with a general anesthesia with the use of rocuronium or vecuronium for endotracheal intubation and maintenance of neuromuscular block;
* Scheduled for surgical procedure in supine position;
* Given written informed consent.

Exclusion Criteria:

* Participants in whom a difficult intubation because of anatomical malformations was expected;
* Is known or suspected to have neuromuscular disorders impairing neuromuscular block (NMB) and/or significant renal dysfunction;
* Is known or suspected to have a (family) history of malignant hyperthermia;
* Is known or suspected to have an allergy to narcotics, muscle relaxants or other medication used during general anesthesia;
* Is receiving medication in a dose and/or at a time point known to interfere with neuromuscular blocking agents such as antibiotics, anticonvulsants and Mg2+;
* Participants in whom the use of neostigmine and/or glycopyrrolate may be contraindicated;
* Had already participated in a sugammadex trial;
* Had participated in another clinical trial, not pre-approved by NV Organon, within 30 days of entering into P05960.
* Females who are pregnant:
* Females of childbearing potential not using any method of birth control: condom or using only hormonal contraception as birth control;
* Females who were breast-feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 198 (Actual)
Dates: Start 2005-11-17 (Actual); Primary Completion 2006-03-06 (Actual); Study Completion 2006-03-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Result] Khuenl-Brady KS, Wattwil M, Vanacker BF, Lora-Tamayo JI, Rietbergen H, Alvarez-Gomez JA. Sugammadex provides faster reversal of vecuronium-induced neuromuscular blockade compared with neostigmine: a multicenter, randomized, controlled trial. Anesth Analg. 2010 Jan 1;110(1):64-73. doi: 10.1213/ane.0b013e3181ac53c3. Epub 2009 Aug 27. PMID 19713265
- [Derived] Blobner M, Eriksson LI, Scholz J, Motsch J, Della Rocca G, Prins ME. Reversal of rocuronium-induced neuromuscular blockade with sugammadex compared with neostigmine during sevoflurane anaesthesia: results of a randomised, controlled trial. Eur J Anaesthesiol. 2010 Oct;27(10):874-81. doi: 10.1097/EJA.0b013e32833d56b7. PMID 20683334
- See also: Click here to access a synopsis of the study results. — http://www.merck.com/clinical-trials/policies-perspectives.html
- Available data/document: CSR Synopsis — http://www.merck.com/clinical-trials/policies-perspectives.html

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants who had a surgical procedure using a general anesthesia of rocuronium or vecuronium for endotracheal intubation and maintenance of neuromuscular block were enrolled in this study.
Groups:
- Rocuronium + Sugammadex: After the last dose of rocuronium, at reappearance of second twitch (T2), a dose of 2.0 mg/kg sugammadex was administered
Period: Overall Study
Arm/Group | Rocuronium + Sugammadex | Rocuronium + Neostigmine | Vecuronium + Sugammadex | Vecuronium + Neostigmine
Started | 49 | 49 | 51 | 49
Treated | 48 | 48 | 48 | 45
Completed | 47 | 47 | 47 | 44
Not Completed | 2 | 2 | 4 | 5
Not completed — Lost to Follow-up | 0 | 1 | 1 | 1
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0
Not completed — Not Treated | 1 | 1 | 3 | 4

BASELINE CHARACTERISTICS:
Population: All Participants As Treated
Groups:
- Total: Total of all reporting groups
Arm/Group | Rocuronium + Sugammadex | Rocuronium + Neostigmine | Vecuronium + Sugammadex | Vecuronium + Neostigmine | Total
Number analyzed (Participants) | 48 | 48 | 48 | 45 | 189
Age, Continuous [Mean (Standard Deviation); unit: Years] | 51 (16) | 48 (14) | 49 (16) | 50 (15) | 49 (15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 24 | 22 | 24 | 87
  Male | 31 | 24 | 26 | 21 | 102
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 9 | 7 | 8 | 29
  Not Hispanic or Latino | 43 | 39 | 41 | 37 | 160
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 0 | 1
  White | 46 | 48 | 48 | 45 | 187
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Time From Start of Administration of Sugammadex or Neostigmine to Recovery of the Fourth Twitch/First Twitch (T4/T1) Ratio to 0.9.
Description: Neuromuscular functioning was monitored by applying repetitive Train-Of-Four (TOF) electrical stimulations to the ulnar nerve every 15 seconds and assessing twitch response at the adductor pollicis muscle. T1 and T4 refer to the amplitudes (heights) of the first and fourth twitches, respectively, after TOF nerve stimulation. The T4/T1 Ratio (expressed as a decimal of up to 1.0) indicates the extent of recovery from neuromuscular blockade (NMB). In this study, twitch responses were recorded until the T4/T1 Ratio reached >= 0.9, the minimum acceptable ratio that indicated recovery from NMB. A faster time to recovery of the T4/T1 Ratio to 0.9 indicates a faster recovery from NMB.
Time Frame: Day 1: From start of sugammadex or neostigmine administration to recovery of T4/T1 ratio to 0.9
Population: All randomized participants who received sugammadex or neostigmine and had at least one efficacy measurement. Imputed recovery times were used in cases of missing times.
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Rocuronium + Sugammadex | Rocuronium + Neostigmine | Vecuronium + Sugammadex | Vecuronium + Neostigmine
Number analyzed (Participants) | 48 | 48 | 48 | 45
Minutes | 1.62 (0.83) | 26.78 (24.60) | 4.47 (9.28) | 23.43 (18.53)

2. Secondary Outcome: Time From Start of Administration of Sugammadex or Neostigmine to Recovery of the T4/T1 Ratio to 0.7
Description: Neuromuscular functioning was monitored by applying repetitive TOF electrical stimulations to the ulnar nerve every 15 seconds and assessing twitch response at the adductor pollicis muscle. T1 and T4 refer to the amplitudes (heights) of the first and fourth twitches, respectively, after TOF nerve stimulation. The T4/T1 Ratio (expressed as a decimal of up to 1.0) indicates the extent of recovery from NMB. A faster time to recovery of the T4/T1 Ratio to 0.7 indicates a faster recovery from NMB.
Time Frame: Day 1: From start of sugammadex or neostigmine administration to recovery of T4/T1 ratio to 0.7
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Rocuronium + Sugammadex | Rocuronium + Neostigmine | Vecuronium + Sugammadex | Vecuronium + Neostigmine
Number analyzed (Participants) | 48 | 48 | 48 | 45
Minutes | 1.17 (0.40) | 9.60 (8.23) | 1.68 (0.57) | 9.52 (10.15)

3. Secondary Outcome: Time From Start of Administration of Sugammadex or Neostigmine to Recovery of the T4/T1 Ratio to 0.8
Description: Neuromuscular functioning was monitored by applying repetitive TOF electrical stimulations to the ulnar nerve every 15 seconds and assessing twitch response at the adductor pollicis muscle. T1 and T4 refer to the amplitudes (heights) of the first and fourth twitches, respectively, after TOF nerve stimulation. The T4/T1 Ratio (expressed as a decimal of up to 1.0) indicates the extent of recovery from NMB. A faster time to recovery of the T4/T1 Ratio to 0.8 indicates a faster recovery from NMB.
Time Frame: Day 1: From start of sugammadex or neostigmine administration to recovery of T4/T1 ratio to 0.8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Rocuronium + Sugammadex | Rocuronium + Neostigmine | Vecuronium + Sugammadex | Vecuronium + Neostigmine
Number analyzed (Participants) | 48 | 48 | 48 | 45
Minutes | 1.32 (0.48) | 15.32 (14.38) | 2.12 (0.87) | 15.33 (13.37)

4. Secondary Outcome: Number of Participants With Clinical Signs of Recovery Assessed by Level of Consciousness, Head Lift and Muscle Weakness, Prior to Transfer to the Recovery Room After Extubation
Description: After anesthesia and prior to transfer to the recovery room after extubation, neuromuscular recovery was assessed by monitoring every 15 minutes the following clinical signs of recovery: level of consciousness (i.e., awake and oriented, arousable with minimal stimulation, responsive only to tactile stimulation); 5-second head lift test (ability to lift the head for 5 seconds); and general muscle weakness
Time Frame: Day 1
Population: All randomized participants who received sugammadex or neostigmine and had at least one efficacy measurement.
Measure: Count of Participants; unit: Participants
Arm/Group | Rocuronium + Sugammadex | Rocuronium + Neostigmine | Vecuronium + Sugammadex | Vecuronium + Neostigmine
Number analyzed (Participants) | 48 | 48 | 48 | 45
Participants
  Consciousness: Awake and oriented | 30 | 35 | 29 | 26
  Consciousness: Arousable with minimal stimulation | 16 | 13 | 17 | 14
  Consciousness: Responsive only to tactile stimuli | 2 | 0 | 2 | 5
  Able to perform the 5 second head lift | 38 | 37 | 40 | 32
  Has general muscle weakness | 3 | 9 | 4 | 6

5. Secondary Outcome: Number of Participants With Clinical Signs of Recovery Assessed by Level of Consciousness, Head Lift and Muscle Weakness, Prior to Discharge From the Recovery Room
Description: Just prior to discharge from the recovery room, neuromuscular recovery was assessed by monitoring every 15 minutes the following clinical signs of recovery: level of consciousness (i.e., awake and oriented, arousable with minimal stimulation, responsive only to tactile stimulation); 5-second head lift test (ability to lift the head for 5 seconds); and general muscle weakness
Time Frame: Day 1
Population: All randomized participants who received sugammadex or neostigmine and had at least one efficacy measurement. One participant from the Rocuronium + Sugammadex treatment group, and one participant from the Vecuronium + Neostigmine treatment group were not analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Rocuronium + Sugammadex | Rocuronium + Neostigmine | Vecuronium + Sugammadex | Vecuronium + Neostigmine
Number analyzed (Participants) | 47 | 48 | 48 | 44
Participants
  Consciousness: Awake and oriented | 46 | 48 | 48 | 43
  Consciousness: Arousable with minimal stimulation | 1 | 0 | 0 | 1
  Consciousness: Responsive only to tactile stimuli | 0 | 0 | 0 | 0
  Able to perform the 5 second head lift | 47 | 48 | 48 | 44
  Has general muscle weakness | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 7 days after sugammadex or neostigmine treatment
Description: All participants as treated
Arm/Group | Rocuronium + Sugammadex | Rocuronium + Neostigmine | Vecuronium + Sugammadex | Vecuronium + Neostigmine
All-Cause Mortality (participants affected / at risk) | 0/48 | 0/48 | 0/48 | 0/45
Serious Adverse Events (participants affected / at risk) | 2/48 | 3/48 | 0/48 | 0/45
Other Adverse Events (participants affected / at risk) | 37/48 | 40/48 | 32/48 | 35/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rocuronium + Sugammadex (N=48) | Rocuronium + Neostigmine (N=48) | Vecuronium + Sugammadex (N=48) | Vecuronium + Neostigmine (N=45)
Subileus (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Postoperative infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Procedural complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Peripheral arterial occlusive disease (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Peripheral ischaemia (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rocuronium + Sugammadex (N=48) | Rocuronium + Neostigmine (N=48) | Vecuronium + Sugammadex (N=48) | Vecuronium + Neostigmine (N=45)
Constipation (Gastrointestinal disorders) | 0 (0) | 6 (6) | 2 (2) | 3 (3)
Dry mouth (Gastrointestinal disorders) | 3 (3) | 5 (5) | 1 (1) | 7 (7)
Nausea (Gastrointestinal disorders) | 12 (13) | 14 (17) | 13 (13) | 16 (19)
Vomiting (Gastrointestinal disorders) | 9 (9) | 6 (6) | 5 (6) | 5 (6)
Chills (General disorders) | 2 (2) | 4 (4) | 4 (4) | 2 (2)
Pain (General disorders) | 11 (12) | 8 (8) | 6 (7) | 5 (5)
Airway complication of anaesthesia (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 1 (2) | 3 (3)
Neuromuscular block prolonged (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Post procedural nausea (Injury, poisoning and procedural complications) | 1 (1) | 3 (3) | 1 (1) | 3 (4)
Post procedural vomiting (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 3 (4)
Procedural complication (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 1 (1) | 4 (5)
Procedural hypertension (Injury, poisoning and procedural complications) | 4 (5) | 3 (3) | 3 (5) | 3 (7)
Procedural hypotension (Injury, poisoning and procedural complications) | 1 (1) | 5 (5) | 0 (0) | 3 (3)
Procedural pain (Injury, poisoning and procedural complications) | 21 (26) | 16 (17) | 18 (21) | 16 (17)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Headache (Nervous system disorders) | 3 (3) | 2 (2) | 3 (3) | 5 (5)
Insomnia (Psychiatric disorders) | 0 (0) | 3 (3) | 1 (1) | 0 (0)
Sleep disorder (Psychiatric disorders) | 2 (2) | 3 (3) | 1 (2) | 1 (1)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 4 (4) | 1 (1) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any scientific paper, presentation, or other communication concerning the clinical trial described in this protocol will first be submitted to the Sponsor, at least six weeks ahead of estimated publication or presentation, for written consent, which shall not be withheld unreasonably.